CLINICAL TRIAL: NCT02570893
Title: A Multicenter, Randomized, Open-label, Phase III Trail of Adjuvant Chemoradiotherapy Versus Adjuvant Radiotherapy in Patients Undergoing Radical Esophagectomy for Pathologic Lymph Node Positive Esophageal Squamous Cell Carcinoma
Brief Title: A Phase III Trail of Adjuvant Chemoradiotherapy Versus Adjuvant Radiotherapy in Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZTOG-1401
Record Dates: First submitted 2015-10-03; First posted 2015-10-07 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Esophageal Cancer
Keywords: Esophageal cancer;adjuvant therapy;chemotherapy;radiotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiotherapy, Adjuvant; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- adjuvant chemoradiotherapy (Experimental): Adjuvant radiotherapy (50.4gray/28fraction) followed by 4 cycles of chemotherapy (Paclitaxel and carboplatin) after radical esophagectomy.
  Interventions: Radiation: Adjuvant radiotherapy; Drug: Paclitaxel and carboplatin
- adjuvant radiotherapy (Experimental): Adjuvant radiotherapy (50.4gray/28fraction) only after radical esophagectomy.
  Interventions: Radiation: Adjuvant radiotherapy

INTERVENTIONS:
Radiation: Adjuvant radiotherapy — Adjuvant radiotherapy (50.4gray/28fraction) followed by 4 cycles of chemotherapy (Paclitaxel and carboplatin) after radical esophagectomy.
  Arms: adjuvant chemoradiotherapy
Radiation: Adjuvant radiotherapy — adjuvant radiotherapy (50.4gray/28fraction) only after radical esophagectomy.
  Arms: adjuvant radiotherapy
Drug: Paclitaxel and carboplatin
  Arms: adjuvant chemoradiotherapy

SUMMARY:
This is a multicenter, randomized, open-label, phase III trail comparing adjuvant chemoradiotherapy (Paclitaxel and carboplatin) to adjuvant radiotherapy in patients undergoing radical esophagectomy for pathologic lymph node positive esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
Patient Population: Age: 18-70y; Thoracic esophageal squamous cell cancer undergoing radical esophagectomy; Clinical stage T1-4, N1-3, M0; Eastern Cooperative Oncology Group (ECOG) score: 0-1; The patients are randomized to 2 arms. Arm A: Adjuvant radiotherapy (50.4gray/28fraction) followed by chemotherapy (Paclitaxel and carboplatin) 4 cycles. Arm B :Adjuvant radiotherapy (50.4gray/28fraction) only

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented squamous cell carcinoma of the thoracic esophagus; undergoing radical esophagectomy; the pathological stage is T(primary tumor)1-4 N(regional lymph nodes)1-3 M(distant metastasis)0 (ESOPHAGUS, Union for International Cancer Control(UICC) 2010) ;
2. Untreated (e.g. radiotherapy, chemotherapy, target therapy and immunotherapy);
3. The expectation of life is more than 6 months;
4. Age: 18~70 years old;
5. Normal hemodynamic indices before the recruitment (including white blood cell count>4.0×109/L, neutrophil count>1.5×109/L, platelet count >100×109/L, hemoglobin≥90g/l, normal liver/kidney function);
6. ECOG (Eastern Cooperative Oncology Group) : 0-1;
7. Able to understand this study and have signed informed consent.

Exclusion Criteria:

1. Have been treated with chemotherapy, radiotherapy and other anti tumor treatment except surgery;
2. Known or suspected of allergy to paclitaxel or carboplatin;
3. Female in pregnancy or lactating;
4. With significant psychological, family, social and other factors which may affect the ability to understand and sign the informed consent;
5. Patients with peripheral neuropathy(CTC grade≥2);
6. With other malignant tumors before the recruitment.
7. The researchers consider that the patient is not appropriate to enroll the study;
8. The patient can't be tolerant to postoperative adjuvant radiotherapy and chemotherapy for serious heart/lung/liver/kidney function, the haematopoietic system diseases, the immune system diseases, the nervous system diseases, cachexia and so on.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
The overall survival | 3 years
  To evaluate the 3 years overall survival of two groups.

SECONDARY OUTCOMES:
Disease-free survival | 3 years
  To evaluate the 3 years disease-free survival of two groups.
Adverse Events | 1 year
  Number and degree of Adverse Events based on Common Toxicity Criteria for Adverse Effects(CTCAE) 4.0
Scores of Quality of life | 1 year
  Assess the quality of life based on FACT-E

CONTACTS AND LOCATIONS:
Overall Officials: Weimin Mao, MD., Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China